CLINICAL TRIAL: NCT03297086
Title: Changes of Angle Kappa After Implantation of Multifocal Intraocular Lenses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Semmelweis University (Other)
Collaborators: Medicontur Kft (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Kappa1
Record Dates: First submitted 2017-09-12; First posted 2017-09-29 (Actual); Last update posted 2017-09-29 (Actual); Status verified 2017-09

CONDITIONS: Cataract; Presbyopia
Keywords: multifocal intraocular lens, angle kappa, presbyopia
MeSH Terms: conditions — Cataract; Presbyopia | interventions — Cataract Extraction

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No

ARMS (2):
- Bi-Flex (Active Comparator): Medicontur Bi-Flex 677MY IOL was implanted into 24 eyes of 12 patients during cataract surgery. Angle kappa, biometric data and IOL decantation were measured.
  Interventions: Procedure: cataract surgery
- ReStor (Active Comparator): and Alcon Acrysof Restor SN6AD1 IOL was implanted into 36 eyes of 18 patients during cataract surgery. Angle kappa, biometric data and IOL decantation were measured.
  Interventions: Procedure: cataract surgery

INTERVENTIONS:
Procedure: cataract surgery — cataract surgery with phacoemulsification and implantation of multifocal posterior chamber intraocular lens

SUMMARY:
The purpose of this study is to evaluate possible changes of angle kappa after multifocal intraocular lens implantation. Presumable influencing factors of postoperative visual axis shift (ie. biometric parameters of the eye) are investigated to determine the degree and direction of angle kappa alterations.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate changes of angle kappa after multifocal intraocular lens implantation.

During cataract surgery Medicontur Bi-Flex 677MY IOL and Alcon Acrysof Restor SN6AD1 IOL are implanted. Optical biometry is carried out for IOL calculation and to measure axial length and angle kappa. Three months after surgery biometry is repeated, IOL position and angle kappa are measured using Scheimpflug-camera.

ELIGIBILITY:
Inclusion Criteria:

* Patients with age related cataract and presbyopia

Exclusion Criteria:

* Patients with previous ocular surgery, trauma, active ocular disease, poorly dilated pupils, or known zonular weakness and corneal astigmatism >1.5 diopters were excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2015-12-01 (Actual); Primary Completion 2016-02-25 (Actual); Study Completion 2017-09-11 (Actual)

PRIMARY OUTCOMES:
Measurement of changes of angle kappa after multifocal intraocular lens implantation. | 3 months
  Changes in magnitude and orientation of angle kappa (deviation between the visual and pupillary axis) are measured before and after cataract surgery with multifoocal intraocular lens implantation. During pre-and postoperative examination optical biometry is carried out using Lenstar LS 900. Optical biometer determines deviation between the visual and pupillary axis that represents angle kappa. Deviation of these axes can be defined by its magnitude and orientation. Location of the pupil centre relative to the visual axis - the reference axis - is determined by x- and y-offsets using trigonometrical analysis.

SECONDARY OUTCOMES:
Determination of influencing effect of biometrical data on postoperative visual axis shift | 3 months
  Biometry data (axial length, keratometry, lens thickness, anterior chamber depth) are measured preoperatively by Lenstar LS 900 optical biometer. Their effect on changes of angle kappa is determined using statistical analysis.
Determination of influencing effect of intraocular lens decentration on postoperative visual axis shift | 3 months
  Three months after cataract surgery postoperative intraocular lens (IOL) position is determined using a rotating Scheimpflug-camera (Galilei G4). IOL decentration is obtained from the distance between the IOL centre and visual axis. The effect of possible IOL decentration on changes of angle kappa is determined using statistical analysis.